CLINICAL TRIAL: NCT06107543
Title: Retrospective Investigation of the Effects of Different Uses of Lidocaine in the Prevention of Hemodynamic Response to Laryngoscopy and Endotracheal Intubation
Brief Title: Lidocaine in the Prevention of Hemodynamic Response to Laryngoscopy and Endotracheal Intubation
Status: Completed | Type: Observational
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Emine Atlı, MD, Anesthesiology and Reanimation, Derince Training and Research Hospital
Other Study IDs: DerinceTRH-EAtli-001
Record Dates: First submitted 2023-09-04; First posted 2023-10-30 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Lidocaine
Keywords: Lidocaine; Intubation; General anaesthesia
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intravenous lidocaine: Patients who received lidocaine intravenously before induction of anesthesia will be considered in this group.
  Interventions: Drug: Iv Lidocaine
- Nebulized lidocaine: Patients who received lidocaine by inhalation with a nebulizer before induction of anesthesia will be considered in this group.
  Interventions: Drug: Nebulized Lidocaine

INTERVENTIONS:
Drug: Nebulized Lidocaine — Before induction of anesthesia, 2% lidocaine + physiological saline was added to a nebulizer and inhaled for 3-5 minutes in the presence of 4-6 liters/minute of oxygen.
  Groups: Nebulized lidocaine
Drug: Iv Lidocaine — Intravenous %2 lidocaine was administered before induction of anesthesia.
  Groups: Intravenous lidocaine

SUMMARY:
Direct laryngoscopy and endotracheal intubation procedure stimulate the sympathetic nervous system, causing catecholamine release into the circulation and consequently hemodynamic changes.There are many studies showing that lidocaine is used intravenously to suppress the sympathetic response to laryngoscopy and endotracheal intubation. Nebulized lidocaine is often used to provide upper airway local anesthesia in fiberoptic guided awake intubation.

In this study, the researchers aimed to compare the results of using intravenous lidocaine and nebulized lidocaine to suppress the hemodynamic response caused by laryngoscopy and endotracheal intubation retrospectively.

Researchers' hypothesis; Nebulized lidocaine administration is more effective than intravenous lidocaine administration in suppressing the hemodynamic response due to laryngoscopy and endotracheal intubation in patients under general anesthesia.

DETAILED DESCRIPTION:
2% lidocaine drug to suppress the hemodynamic response due to laryngoscopy and endotracheal intubation; patients administered intravenously will be evaluated in one group, and patients administered inhaled through a nebulizer will be evaluated in another group.

Nebulized lidocaine in the researchers' clinic; it is administered by adding 2% lidocaine + physiological saline to a nebulizer and inhaling for 3-5 minutes in the presence of 4-6 liters/minute of oxygen.

Preoperative examination forms and intraoperative follow-up forms of the patients included in the study will be examined by the researchers. The dose of lidocaine applied and the method of administration will be recorded. In addition, the agents used in anesthesia induction (fentanyl, propofol, rocuronium bromide, etc.) and the hemodynamic changes of the patients (heart rate, systolic blood pressure, diastolic blood pressure, mean arterial pressure,oxygen saturation) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 and under the age of 80 who underwent surgery under general anesthesia

Exclusion Criteria:

* Patients under the age of 18 and over the age of 80
* Patients who are not operated under general anesthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 80 patients over the age of 18 and under the age of 80 who underwent surgery under general anesthesia in the operating room will be included in the study.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-22 (Actual)

PRIMARY OUTCOMES:
Heart Rate | Just before induction of anesthesia
  Patients were monitored with a three-lead ECG in the operating room and their heart rates were recorded as beats per minute. (.../min)
Heart Rate | Immediately after induction of anesthesia
  Patients were monitored with a three-lead ECG in the operating room and their heart rates were recorded as beats per minute. (.../min)
Heart Rate | 5 minutes and 10 minutes after direct laryngoscopy and endotracheal intubation
  Patients were monitored with a three-lead ECG in the operating room and their heart rates were recorded as beats per minute. (.../min)
Blood Pressure | Just before induction of anesthesia
  The patients were monitored in the operating room by wearing a noninvasive blood pressure cuff and measurements were taken at 5-minute intervals. Systolic blood pressure, diastolic blood pressure and mean arterial pressure were recorded in mmHg.
Blood Pressure | Immediately after induction of anesthesia
  The patients were monitored in the operating room by wearing a noninvasive blood pressure cuff and measurements were taken at 5-minute intervals. Systolic blood pressure, diastolic blood pressure and mean arterial pressure were recorded in mmHg.
Blood Pressure | 5 minutes and 10 minutes after direct laryngoscopy and endotracheal intubation
  The patients were monitored in the operating room by wearing a noninvasive blood pressure cuff and measurements were taken at 5-minute intervals. Systolic blood pressure, diastolic blood pressure and mean arterial pressure were recorded in mmHg.
Oxygen Saturation | Just before induction of anesthesia
  The patients were monitored with a pulse oximetry device in the operating room and their oxygen saturation % (spO2) was recorded.
Oxygen Saturation | Immediately after induction of anesthesia
  The patients were monitored with a pulse oximetry device in the operating room and their oxygen saturation % (spO2) was recorded.
Oxygen Saturation | 5 minutes and 10 minutes after direct laryngoscopy and endotracheal intubation
  The patients were monitored with a pulse oximetry device in the operating room and their oxygen saturation % (spO2) was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Derince Training and Research Hospital, Kocaeli, Turkey (Türkiye)

REFERENCES:
- [Result] Baronia AK, Singh PK, Maheshwari A, Jain VK, Mittal P, Pant KC. Inhaled lidocaine for prevention of hemodynamic changes in laryngoscopy and intubation. J Neurosurg Anesthesiol. 1992 Jul;4(3):154-9. doi: 10.1097/00008506-199207000-00002. PMID 15815458
- [Result] Sklar BZ, Lurie S, Ezri T, Krichelli D, Savir I, Soroker D. Lidocaine inhalation attenuates the circulatory response to laryngoscopy and endotracheal intubation. J Clin Anesth. 1992 Sep-Oct;4(5):382-5. doi: 10.1016/0952-8180(92)90160-3. PMID 1389192